CLINICAL TRIAL: NCT05862077
Title: Long-term Exercise Effect of EX1 Exercise Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Samsung Electronics (Industry)
Responsible Party: Principal Investigator, Yun-Hee Kim, Dr., Ph.D., Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2023-03-005
Record Dates: First submitted 2023-03-22; First posted 2023-05-17 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Aging
Keywords: Exercise program; Wearable hip assist robot; Gait

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Overground walking exercise without EX1 (Sham Comparator): Exercise consists of 30 minutes of overground walking.
  Interventions: Device: Without Wearable Hip Assist Robot(EX1)
- Exercise program 1 with EX1 (Experimental): Exercise program 1 consists of 30 minutes of overground walking.
  Interventions: Device: Wearable Hip Assist Robot(EX1); Behavioral: Exercise Program 1
- Exercise program 2 with EX1 (Experimental): Exercise program 2 consists of 30 minutes of overground walking.
  Interventions: Device: Wearable Hip Assist Robot(EX1); Behavioral: Exercise Program 2

INTERVENTIONS:
Device: Wearable Hip Assist Robot(EX1) — EX1 is a hip-type assist device developed by Samsung Electronics.
  Arms: Exercise program 1 with EX1; Exercise program 2 with EX1
Behavioral: Exercise Program 1 — Exercise program 1 for fast walking by applying resistance and assist mode of EX1
  Arms: Exercise program 1 with EX1
Behavioral: Exercise Program 2 — Exercise program 2 for normal walking by applying resistance and assist mode of EX1
  Arms: Exercise program 2 with EX1
Device: Without Wearable Hip Assist Robot(EX1) — Overground walking without EX1
  Arms: Overground walking exercise without EX1

SUMMARY:
The purpose of this study was to investigate the effect of a long-term exercise program using a wearable exoskeleton robot (EX1) on muscular strength in healthy adults aged 19 to under 65 years, compared to an exercise program without EX1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 19 to less than 65 years without a history of central nervous system disease

Exclusion Criteria:

* Those who have difficulty walking independently due to problems such as visual field defects or fractures
* Those who have difficulty participating in exercise programs due to adult diseases such as uncontrolled hypertension and diabetes
* Those who are at risk of falling while walking due to severe dizziness
* Those who are less than 140 cm or more than 185 cm in height that is not suitable size for the wearing of the walking assistance robot
* Those who are overweight based on body mass index (BMI) 35 or higher

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Change on gait function (muscle activation) | Session 0 (initial visit); after session 18 (at approximately 6 weeks)
  All subjects perform overground walking to assess the change of muscle activation after the interventions using a surface EMG (6 channels).

SECONDARY OUTCOMES:
Change in heart rate | Every session (total 18 sessions/ 30 minutes)
  All subjects are measured for heart rate during the intervention.
Reduction in stress level | Session 0 (initial visit); after session 18 (at approximately 6 weeks)
  We evaluate the subject's usual stress level through a questionnaire. The Perceived Stress Scale (PSS-10) is a 10-item questionnaire originally developed by Cohen et al. (1983) widely used to assess stress levels in young people and adults.
  The questions ask about feelings and thoughts during the last month. In each case, respondents are asked how often they felt a certain way on a five-point scale from 'never' to 'very often'. Answers are then scored as follow: Never = 0; Almost never = 1; Sometimes = 2; Fairly often = 3; Very often = 4.
  The PSS score is then obtained by summing across all items. Higher scores indicate higher levels of perceived stress.
Reduction in body fat percentage | Session 0 (initial visit); after session 18 (at approximately 6 weeks)
  All subjects are measured for body fat before and after the intervention.
User Satisfaction Questionnaire | After session 18 (at approximately 6 weeks)
  We evaluate the satisfaction questionnaire for EX1 use and exercise program.
Change on gait function (kinematic) | Session 0 (initial visit); after session 18 (at approximately 6 weeks)
  All subjects perform overground walking to assess the change of kinematic using a motion analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Sungkyunkwan University, Suwon, South Korea

REFERENCES:
- [Derived] Lee SH, Kim E, Kim J, Kim D, Lee D, Lee HJ, Kim YH. Effect of Programed Walking Exercise Using Bot Fit in Younger Adults. Sports Med Open. 2024 Oct 14;10(1):112. doi: 10.1186/s40798-024-00773-x. PMID 39400778